CLINICAL TRIAL: NCT06788457
Title: Assessment and Validation of a Device for Measuring Hydrogen Peroxide in Exhaled Breath Condensate in Healthy Volunteers
Brief Title: Measuring Hydrogen Peroxide in Exhaled Breath Condensate in COPD
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21IC7212
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Proof of Concept Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Exhaled breath condensate (EBC)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Healthy individuals, free of significant disease.
  Interventions: Device: Exhaled Breath Condensate
- Participants with COPD: A diagnosis of COPD.
  Interventions: Device: Exhaled Breath Condensate

INTERVENTIONS:
Device: Exhaled Breath Condensate — Measurement of hydrogen peroxide in exhaled breath

SUMMARY:
Following a successful pilot study and a clinical assessment in healthy volunteers (ClinicalTrials.gov ID: NCT05844553) this study aims to evaluate the accuracy and precision of an Exhaled Breath Condensate (EBC) device in patients with COPD. The study will evaluate the reproducibility of 3 measurements a month apart in real breath samples. This will take place at the Clinical Research Facility (CRF) at the Royal Brompton Hospital. Real biological specimens are complex and there is the potential for losses of precision and accuracy. This can only be evaluated by comparison with established methodology. Secondly, whilst many reports can correctly classify COPD patients, there are substantial variations in absolute levels between researchers. It has been shown with artificial samples that correcting for variations in heat and mass transport can substantially reduce these variations. Collecting replicate samples from patients with COPD will allow the evaluation within this patient group.

DETAILED DESCRIPTION:
The study aim is to recruit 15 patients with COPD and 15 healthy volunteers in order tevaluate the analytical performance of the device and the data processing and consistency of measurements over a 3-month period.

Three successive measurements will be made at monthly intervals in each patient with COPD and with each healthy volunteer requiring them to visit the Hospital on three occasions. The first visit also includes screening which will take up to 1 hour.

Firstly, each potential participant will be sent a participant information sheet.

If they decide that they wish to take part in the research study, they will be asked to come to the Clinical Research Facility (CRF) at the Royal Brompton Hospital, for screening where the research team will further explain the study to the participant. A hard copy of the participant information sheet will be provided at the appointment and participants will be encouraged to ask questions. Participants will then be presented with a consent form which they will be asked to sign before any procedures are made.

ELIGIBILITY:
Inclusion Criteria:

COPD participants:

* A diagnosis of COPD.
* Not current smokers
* Stable COPD (no chest infection requiring antibiotics and/or oral steroids in the past 1 month).
* Able to give written informed consent prior to participation in the study including all of its procedures.
* Male or female subject aged 18 years and above at screening.
* Able to complete the study and all measurements.
* Able to read, comprehend, and write at a sufficient level to complete study related materials

Healthy subjects:

* non-smokers
* Healthy individuals, free of significant disease.
* Able to give written informed consent prior to participation in the study including all of its procedures.
* Able to comply with the requirements and restrictions listed in the consent form.
* Male or female subject aged 18 years and above at screening.
* Able to complete the study and all measurements.
* Able to read, comprehend, and write at a sufficient level to complete study related materials.

Exclusion Criteria:

COPD Participants:

* We will not recruit subjects who lack the capacity to consent.
* Current or past diagnosis of asthma.
* History of any chronic respiratory diseases other than COPD.
* History of another medical condition, which in the opinion of the Unit Physician, contraindicates his/her participation in the study.

Unstable respiratory disease in the last four weeks prior to the screening visit (indicated by any change in their maintenance inhaled therapy or who have had a lower respiratory tract infection in the previous four weeks).

* Evidence of a respiratory exacerbation requiring emergency room treatment and/or hospitalisation within four weeks before screening.
* Use of systemic (oral or intravenous) steroids 4 weeks prior to inclusion (injectable depot steroids 6 weeks) or more than 3 periods during the last 12 months.
* Patients who have evidence of alcohol or substance abuse.
* Participation in another clinical trial with an investigational drug in the four weeks preceding the screening visit.
* Those, in the opinion of the investigator, who may prove non-compliant with study procedures.
* History of an upper or lower respiratory infection (including coryza) within 3 weeks of baseline assessments (assessments and entry could be deferred.

Healthy subjects:

* A history of recreational drug use or allergy which in the opinion of the investigators contra-indicates their participation.
* Participation within 3 months in any other study testing a new molecular entity or drug or involving invasive procedures.
* Those, in the opinion of the investigator, who may prove non-compliant with study procedures.
* History of an upper or lower respiratory infection (including coryza) within 3 weeks of baseline assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with COPD and Heathy participants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Precision and accuracy of the EBC device in COPD & healthy participants. | 12 months
  This will be assessed by comparison with the gold standard fluorometry and mass spectrometry methods.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Usmani, MBBS, MRCP, PhD, Principal Investigator — Imperial College London
Locations (1):
- Clinical Research Facility, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT06788457/Prot_000.pdf